CLINICAL TRIAL: NCT04221581
Title: Prospective Observational Clinical Study Conducted on Patient Operated With a Total Knee Prosthesis FHK ASYMETRIQUE to Confirm Security and Performance of the Device Over a Period of 10 Years
Brief Title: Study Conducted on Patients Operated With a FHK ASYMETRIQUE to Confirm Security and Performance of the Device
Status: Active, not recruiting | Type: Observational
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-38
Record Dates: First submitted 2019-12-18; First posted 2020-01-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Knee Disease
Keywords: Knee; Arthroplasty; Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving FHK ASYMETRIQUE prosthesis
  Interventions: Device: Knee prosthesis - FHK ASYMETRIQUE total knee prosthesis

INTERVENTIONS:
Device: Knee prosthesis - FHK ASYMETRIQUE total knee prosthesis — FHK ASYMETRIQUE prosthesis are intended to be implanted in the tibial and femoral regions during total knee arthroplasty in order to restore joint function.

SUMMARY:
This study is a post-market clinical follow-up conducted in order to collect long-term data on security and performance of the FHK asymetrique prosthesis, which is intended to be implanted in case of total knee replacement, when used in real life conditions according to the instructions for use.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the security of the FHK ASYMETRIQUE prosthesis by calculating the survival rate up to 10 years of follow-up.

The secondary objectives are to evaluate the security and performance of the device by assessing radiological data, gathering complications and evaluating functional score up to 10 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults subjects (≥18 years old).
* Subject implanted with FHK ASYMETRIQUE prosthesis in one of the following indication according to the instructions for use: knee disorders; Aseptic condylar necrosis.
* Subject who received an information form and is willing to participate in the study.

Exclusion Criteria:

* Contraindications described in the instructions for use
* Usual surgical contraindications
* Patients objecting to participate in this study
* Subject who is not able to express his/her non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from participating hospitals will be enrolled as part of their clinical routine care
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2034-01-22 (Estimated); Study Completion 2034-01-22 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | 10 years post-op
  Survival rate

SECONDARY OUTCOMES:
Radiological evaluation | preoperative, 3 months post-op, 1 year post-op, 3 years post-op, 5 years post-op, 10 years post-op
  Radiological results such as stability, osteointegration will be evaluated. The HKA angle will be measured. It is the angle (in degrees) between the center of the femoral head, the center of the knee and the center of the tibio-fibular mortise. This radiological evaluation is a usual assessment used in the follow-up of patients operated for a total knee replacement.
Rate of complications | peroperative, 3 months postoperative, 1 year post-op, 3 years post-op, 5 years post-op, 10 years post-op
  All complications will be gathered during intervention and up to 10 years postoperatively.
Functional outcomes such as pain, mobility. | preoperative, 3 months post-op, 1 year post-op, 3 years post-op, 5 years post-op, 10 years post-op
  Functional outcomes will be determined by the IKS score. New IKS score range from 0 to 200 with a physical score on 100 points (pain, knee's mobility, abnormal laxity, flexion deformity and Hips knee Ankle) and a functional score on 100 points (walking distance, difficulty with stairs and use of walking aids).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Pasteur, Colmar
  - Clinique Mutualiste de la Porte de l'Orient, Lorient
  - Médipôle Garonne, Toulouse

IPD SHARING:
Plan to Share IPD: No